CLINICAL TRIAL: NCT03143049
Title: Randomized Phase 3 Study of Pomalidomide-Cyclophosphamide-Dexamethasone (PCD) Versus Pomalidomide-Dexamethasone (PD) in Relapse or Refractory Myeloma. An AMN Study
Brief Title: Pomalidomide-Cyclophosphamide-Dexamethasone (PCD) Versus Pomalidomide-Dexamethasone (PD) in Relapse or Refractory Myeloma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Celgene (Industry); International Myeloma Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMN003
Record Dates: First submitted 2017-04-13; First posted 2017-05-08 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-03

CONDITIONS: Relapse Multiple Myeloma
Keywords: Pomalidomide

STUDY DESIGN:
Intervention Model Description: This is a randomised phase 3 study in Asian patients with relapse multiple myeloma after prior bortezomib and lenalidomide who will be treated by PD or PCD. Randomisation will be 1:1 using a computer algorithm. There will be no blinding. The patient in the 2 arms will be stratified according to ISS stage 1 or 2 versus stage 3.
  Cross-over for patients randomised to Pomalidomide and Dexamethasone at progression:
  Upon progression, patients randomized to pomalidomide and dexamethasone (PD) can cross-over to the PCD arm and have cyclophosphamide added to their regimen according to the PCD regimen. Cyclophosphamide should be added at the beginning of a cycle. They can continue on PCD until further progression. However for these PD patients that cross-over to PCD, the primary endpoint for analysis will be based on response and progression on PD.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pomalidomide, Cyclophosphamide, Dex (PCD) (Experimental)
  Interventions: Drug: PCD
- Pomalidomide, Dex (PD) (Active Comparator)
  Interventions: Drug: PD

INTERVENTIONS:
Drug: PCD — For PCD, patients will be treated as follows: PO pomalidomide 4mg from D1-21, PO cyclophosphamide 400mg on D1, 8 and 15, and PO or IV dexamethasone 40mg D1, 8, 15 and 22 in a 28-day cycle.
  Patients will be assessed every 28 days (+/- 10 days). Patients shall receive the treatment until disease progression, unacceptable toxicity as determined by treating physician, withdrawal of consent or mortality (whichever occurs first).
  Arms: Pomalidomide, Cyclophosphamide, Dex (PCD)
Drug: PD — For PD, Patients will be treated as follows: PO pomalidomide 4mg from D1-21 and PO or IV dexamethasone 40mg D1, 8, 15 and 22 in a 28-day cycle.
  Patients will be assessed every 28 days (+/- 10 days). Patients shall receive the treatment until disease progression, unacceptable toxicity as determined by treating physician, withdrawal of consent or mortality (whichever occurs first).
  Arms: Pomalidomide, Dex (PD)

SUMMARY:
Myeloma patients who relapse after prior treatment with bortezomib and lenalidomide have survival of less than 1 year. Recently, a randomized study of Pomalidomide and dexamethasone conducted in compared with placebo and dexamethasone showed that pomalidomide can improve survival of this group of patients. As a result, pomalidomide is now approved by the FDA and EMA for use in patients with relapsed/refractory myeloma previously treated with bortezomib and lenalidomide. We have conducted a study using Pomalidomide plus Dexamethasone (PD) in Asian patients, which showed good efficacy and safety profile. More important for patients with suboptimal response to PD will achieve a clinically meaningful response with the addition of oral cyclophosphamide (PCD). In the United States, a small randomised phase 2 study of PCD versus PD showed that PCD have a higher response rates, produce deeper response and correspondingly longer progression free survival. There is till date no randomised phase 3 study between these regimens. This will be important to determine what is the best combination including pomalidomide for use in relapse myeloma.

DETAILED DESCRIPTION:
In this study, we will prospectively enrol 120 Asian patients with relapsed myeloma after prior treatment with bortezomib and lenalidomide, and randomised them between PCD and PD (60 in each arms). Centers in Singapore, Korea, Taiwan, and Hong Kong will participate in this study.

Pomalidomide is a new immunomodulatory drug, which has been shown to be active in myeloma patients who relapse after bortezomib and lenalidomide. A recent phase III study comparing pomalidomide plus dexamethasone with placebo plus high dose dexamethasone in patients with prior exposure to bortezomib and lenalidomide, showed that the use of pomalidomide significantly improve the overall survival of these patients. In an Asian study, it appears that the addition of cyclophosphamide can induce further response in patients without a response to PD. In the United States, a small randomised phase 2 study of PCD versus PD showed that PCD have a higher response rates, produce deeper response and correspondingly longer progression free survival. Our hypothesis is therefore that PCD will be better than PD and should be the standard pomalidomide containing regimen for relapse myeloma patients. This combination will also be highly relevant to Asian patients because cyclophosphamide is a relatively cheap drug and the combination will be cost effective if proven to be better than PD.

Rationale for the Study Purpose There is a relative lack of data on the efficacy and tolerability of PCD in Asian Patients. The current study will also allow us to test if PCD is better than PD in the treatment of relapse myeloma patients.

Rationale for Study Population The study population will be myeloma patients who have relapsed following prior treatment with bortezomib and lenalidomide. Pomalidomide is the current approved treatment choice for this group of patients and a common indication for us in Asia.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple myeloma, diagnosed according to standard criteria, with relapsing and refractory disease at study entry
2. Patients must have evaluable multiple myeloma with at least one of the following (within 21 days of starting treatment)

   1. Serum M-protein ≥ 0.5g/dL, or
   2. In subjects without detectable serum M-protein, Urine M-protein ≥ 200mg/24 hour, or serum free light chai (sFLC) > 100mg/L (involved light chain) and an abnormal kappa/Lambda ratio
3. Can receive up to 6 lines of prior treatment. (Induction therapy followed by stem cell transplantation and consolidation/maintenance therapy will be considered as one line of treatment)
4. Must be relapse refractory to prior lenalidomide and bortezomib. Refractoriness is defined as disease progression on treatment or progression within 6 months after the last dose of a given therapy. Relapse is defined according to the criteria of IMWG
5. Males and females ≥ 18 years of age or > country's legal age for adult consent
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
7. Patients must meet the following clinical laboratory criteria with 21 days of starting treatment:

   1. Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet ≥ 50,000/mm3 (≥ 30,000/mm3 if myeloma involvement in the bone marrow is >50%)
   2. Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
   3. Calculated creatinine clearance ≥ 30mL/min or creatinine < 3mg/dL.
8. Female patients who:

   1. Are naturally postmenopausal for at least 2 year before enrolment
   2. Are surgically sterile
   3. If they are of childbearing potential**, agree to

      * adhere to the pomalidomide pregnancy prevention risk management program in Appendix 8 :
      * All women of childbearing potential must agree to have two negative pregnancy test within 10-14 days and 24hrs before commencing pomalidomide and use two reliable methods of contraception simultaneously or practice complete abstinence from any heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study; 2) while participating in the study; 3) dose interruptions; and 4) for at least 28 days after study treatment discontinuation. The two methods of reliable contraception must include one highly effective method and one additional effective method to prevent pregnancy, not plan on conceiving children during or within 6 months following pomalidomide. (See Appendix 8 Pregnancy Prevention and Risk Management Program)
9. Male patients, even if surgically sterilized (i.e. status post-vasectomy), who:

   1. Agree to practice effective barrier contraception during the entire study treatment period and through 28 days after the last dose of study treatment, OR
   2. Agree to completely abstain from heterosexual intercourse, AND
   3. Must also adhere to the guidelines of the pomalidomide pregnancy prevention and risk management program
10. Written informed consent in accordance with federal, local and institutional guidelines

    * A female of childbearing potential (FCBP) is defined as a sexually mature woman who: 1 has not undergone a hysterectomy or bilateral oophorectomy or 2, has not been naturally post-menopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (I.E, has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

1. Female patients who are lactating or pregnant
2. Multiple Myeloma of IgM subtype
3. Glucocorticoid therapy (prednisolone > 30mg/day or equivalent) within 14 days prior to informed consent obtained
4. POEMS syndrome
5. Plasma cell leukemia or circulating plasma cells ≥ 2 x 109/L
6. Waldenstrom's Macroglobulinaemia
7. Patients with known amyloidosis
8. Chemotherapy with approved or investigation anticancer therapeutics within 21 days prior to starting pomalidomide treatment
9. Focal radiation therapy within 7 days prior to start of pomalidomide. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to start of pomalidomide
10. Immunotherapy (excluding steroids) 21 days prior to start of pomalidomide
11. Major surgery (excluding kyphoplasty) within 28 days prior to start of pomalidomide
12. Active congestive heart failure (New York Heart Association [NYHA] Class III or IV), symptomatic ischaemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within 4 months prior to informed consent obtained
13. Known HIV seropositive, hepatitis C infection, and/or hepatitis B (except for patients with hepatitis B surface antigen or core antibody receiving and responding to antiviral therapy directed at hepatitis B: these patients are allowed)
14. Patients with known cirrhosis
15. Second malignancy within the past 3 years except:

    1. Adequately treated basal cell or squamous cell skin cancer
    2. Carcinoma in situ of the cervix
    3. Breast carcinoma in situ with full surgical resection
16. Patients with myelodysplastic syndrome
17. Patients with steroid or lenalidomide hypersensitivity
18. Prior treatment with pomalidomide
19. Ongoing graft-versus-host disease
20. Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to starting pomalidomide treatment
21. Contraindication to any of the required concomitant drugs or supportive treatments
22. Any clinically significant medical disease or psychiatric condition that, in the investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Assessed up to 100 months
  Defined as the time from commencement of treatment with either PCD or PD to disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Assessed up to 100 months
  Defined as the percentage of patients enrolled that achieve a complete response (CR), or stringent complete response (sCR), or very good partial response (VGPR), or partial response (PR) based on the International Myeloma Working Group criteria anytime from commencement of treatment to the end of study.
Overall survival (OS) | An average of 5 years
  Defined as the time from commencement of treatment to the date of death
Duration of response (DOR) | Assessed up to 100 months
  Defined as the time from first evidence of PR or VGPR, or CR, or sCR to confirmation of disease progression or death due to any cause.
Number of Participants affected by Adverse Events | From the time of enrolment into study till 3 years from the date of the last patient randomized
  Assessed on the basis of the frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wee Joo Chng, Principal Investigator — National University Hospital, Singapore
Locations (5):
- Queen Mary Hospital, Hong Kong, Hong Kong
- Japan, Japan
- National University Hospital, Singapore, Singapore
- South Korea, South Korea
- National Taiwan University, Taipei, Taiwan

REFERENCES:
- [Background] Miguel JS, Weisel K, Moreau P, Lacy M, Song K, Delforge M, Karlin L, Goldschmidt H, Banos A, Oriol A, Alegre A, Chen C, Cavo M, Garderet L, Ivanova V, Martinez-Lopez J, Belch A, Palumbo A, Schey S, Sonneveld P, Yu X, Sternas L, Jacques C, Zaki M, Dimopoulos M. Pomalidomide plus low-dose dexamethasone versus high-dose dexamethasone alone for patients with relapsed and refractory multiple myeloma (MM-003): a randomised, open-label, phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1055-1066. doi: 10.1016/S1470-2045(13)70380-2. Epub 2013 Sep 3. PMID 24007748
- [Background] Larocca A, Montefusco V, Bringhen S, Rossi D, Crippa C, Mina R, Galli M, Marcatti M, La Verde G, Giuliani N, Magarotto V, Guglielmelli T, Rota-Scalabrini D, Omede P, Santagostino A, Baldi I, Carella AM, Boccadoro M, Corradini P, Palumbo A. Pomalidomide, cyclophosphamide, and prednisone for relapsed/refractory multiple myeloma: a multicenter phase 1/2 open-label study. Blood. 2013 Oct 17;122(16):2799-806. doi: 10.1182/blood-2013-03-488676. Epub 2013 Aug 16. PMID 23954889
- [Derived] Kim JS, Song Y, Jen WY, Chim CS, Lee JJ, Yoon SS, Ng SC, Gan GG, Handa H, Lee JH, Kim K, Ito S, Huang JS, Min CK, Ooi Gaik Ming M, de Mel S, Soekojo C, Li X, Awasthi N, Pokharkar Y, Durie BG, Chng WJ. Randomized Phase 3 study of pomalidomide cyclophosphamide dexamethasone versus pomalidomide dexamethasone in relapse or refractory myeloma: an Asian Myeloma Network study (AMN003). Blood Cancer J. 2025 Oct 6;15(1):155. doi: 10.1038/s41408-025-01356-z. PMID 41052983